CLINICAL TRIAL: NCT00768677
Title: Open-Label Study of Topiramate for Binge Eating Disorder and Bulimia Nervosa Among Adolescents
Brief Title: Topiramate for Binge Eating Disorder Among Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Zucker Hillside Hospital (Other)
Responsible Party: Ema Saito, The Zucker Hillside Hospital
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 03-04-063
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2008-10-08 (Estimated); Status verified 2008-09

CONDITIONS: Eating Disorders; Bulimia Nervosa
Keywords: binge eating behavior; adolescents
MeSH Terms: conditions — Feeding and Eating Disorders; Bulimia Nervosa; Binge-Eating Disorder | interventions — Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: topiramate

SUMMARY:
This is a study of topiramate to see whether topiramate decreases binge eating behavior among adolescents and young adults. The investigators did also checked whether topiramate affected cognitive function or not.

ELIGIBILITY:
Inclusion Criteria:

Subjects (aged 12 to 23) were included if they

* Met the criteria of bulimia nervosa or eating disorder NOS with binge-eating behavior in DSM-IV-TR,
* Had weight > or = 100th % of expected body weight for their age,
* Engaged in binge eating at least once a week for 9 out of the 12 weeks prior to the study entry, and
* Were judged by a clinician to be stable enough to be treated for their psychiatric condition as an outpatient (i.e, no acute suicidality, hallucination, unstable vital signs or persistently abnormal laboratory results due to eating disorder).

Exclusion Criteria:

* Subjects whose psychotropic medications had been changed within 4 weeks prior to the entry or who had started psychotherapy within 3 months prior to the entry were excluded.
* Subjects were also excluded if they were taking carbonic anhydrase inhibitors, carbamazepine, phenytoin, phenobarbital, valproic acid, evening primrose oil or oral contraceptives.
* Other exclusion criteria were: history of substance use disorders within the 6 months prior to study, IQ < or = 70, medical conditions causing weight loss (i.e., hyperthyroidism, diabetes mellitus type 1, malignancy) or that contra indicate treatment with topiramate (nephrolithiasis or glaucoma), history of non response or poor tolerance to topiramate in the past and history of non-adherence to medication treatment.

Ages: 12 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2003-07

CONTACTS AND LOCATIONS:
Locations (1):
- The Zucker Hillside Hospital, Glen Oaks, New York, United States